CLINICAL TRIAL: NCT06600984
Title: Efficacy of Whole Body Vibration on Fascicle Length and Joint Angle in Children With Hemiplegic Cerebral Palsy
Brief Title: WBV on Fascicle Lenght and Knee Joint Angle in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associated professor of pediatric physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004996
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Fascicle length; Hemiplegia; Range of motion; Whole body vibration
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy group (Experimental): Control group: received a designed physical therapy program
  Interventions: Other: designed physiotherapy program
- whole body vibration group (Experimental): experimental group: received a designed physical therapy program in addition to WBV for 12 weeks
  Interventions: Device: whole body vibration; Other: designed physiotherapy program

INTERVENTIONS:
Device: whole body vibration — On a vibration platform, the children went into a complete squat. The device was calibrated at a frequency of 30 Hz, an amplitude of 2 mm, and a duration of 5 minutes. After the vibration was turned on, the children were told to stay in the squatting position and to report any discomfort that could occur. The vibration automatically shut off after five minutes. The children then rested for a minute. Next, under the identical conditions as for the squatting position, they were instructed to stand on the vibration platform for five minutes with the therapist's assistance. Consequently, WBV was applied for a total of 10 minutes during each session.
  Other Names: WBV
  Arms: whole body vibration group
Other: designed physiotherapy program — structured therapeutic exercise program that included neurodevelopmental approaches, balance exercises, milestone facilitation, stretching exercises, and postural reaction facilitation. The program was conducted for one hour each day, three days a week.
  Other Names: physical therapy program

SUMMARY:
This study investigates the effects of WBV on fascicle length, knee joint angle and function in children with spastic hemiplegic cerebral palsy

DETAILED DESCRIPTION:
to study the effect of WBV on fascicle length, knee joint angle and function in children with spastic hemiplegic cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* Ages varied from four to six years of both sex
* hemiplegic CP children, were suffering from knee joint flexion deformity due to hamstring muscles tightness
* Level I and II motor function, according to the Growth Motor Function Classification System (GMFC) expanded and revised
* Degree of spasticity ranged from 1 to 2 according to modified Ashworth scale
* All children received neuro-developmental techniques

Exclusion Criteria:

* Other causes of knee flexion deformities
* Previous history of orthopedic surgery in knee joint
* Visual or auditory problems
* Seizures
* Sensory or perceptual deficits
* Any acute illness at the time of collection of data.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Knee range of motion | 12 weeks
  Each child in both groups had their knee joint's extension angle measured before and after a 12-week therapy program began using an absolute + AxisTM Digital Goniometer
Fascicle length of hamstring muscle | 12 weeks
  The biceps femoris muscle's muscle fascicle length was measured at a frequency of 7.5 MHz using GE LOGIQ P6 ultrasonography equipment
gross motor function | 12 weeks
  Gross Motor Functional Measurement-88 : is a common principle-test designed to assess changes in function in various milestones for children with cerebral palsy 0 = does not initiate
  1. = initiates
  2. = partially completes
  3. = completes

CONTACTS AND LOCATIONS:
Locations (1):
- mostafa ALI, Giza, Married, Egypt

IPD SHARING:
Plan to Share IPD: No